CLINICAL TRIAL: NCT04528602
Title: The Effect of Diaper Change Position on Neonatal Comfort and Heart Rate, Respiratory Rate and Oxygen Saturation in Preterm Infants
Brief Title: The Effect of Diaper Change Position on Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-5/12
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Infant, Premature, Diseases
Keywords: preterm; diaper change; comfort; position
MeSH Terms: conditions — Infant, Premature, Diseases; Premature Birth | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Extended leg position) Group (Experimental): In the control (Extended leg position) group of the study, diaper change will be performed after the legs of the babies are brought to extension.
  Interventions: Procedure: Control (Extended leg position) Group
- Experimental (Legs are flexed toward abdomen) Group (Experimental): In the experimental (Legs are flexed toward abdomen) group, the diaper change will be performed after the legs of the babies are brought closer to the abdomen while maintaining their flexion leg position.
  Interventions: Procedure: Experimental (Legs are flexed toward abdomen) Group

INTERVENTIONS:
Procedure: Control (Extended leg position) Group — Common procedure steps -Legal representatives of the infants will sign an informed consent form. Materials (soap, napkin, non-sterile gloves, diaper, wet cotton towels for newborns, waste container, diaper change mat) will be prepared.
  Hands will be washed and gloves will be worn. Tapes of the infant's dirty diaper will be opened.
  For the Control Group
  -The infant will be grasped on the legs, the legs will be given extension position and lifted up.
  The dirty diaper will be folded in two and the perineum area will be wiped with a wet cotton towel from the front to the back.
  The infant's feet will be freed. The dirty diaper will be removed and thrown into the general waste bin. The used gloves will be removed.
  The infant's legs will be given in extension position and a clean diaper will be placed under them.
  Tapes of the clean diaper will be fastened. Hands will be washed after the procedure Data will be collected before, during, after and 3 minutes after application.
  Arms: Control (Extended leg position) Group
Procedure: Experimental (Legs are flexed toward abdomen) Group — Procedure steps for the Experimental Group
  * Common procedure steps
  * The infant will be grasped on the legs; the legs will be kept in the flexion position and approached toward the abdomen.
  * The dirty diaper will be folded in two and the perineum area will be wiped with a wet cotton towel from the front to the back.
  * The infant's feet will be freed.
  * The dirty diaper will be removed and thrown into the general waste bin. The used gloves will be removed and thrown into the medical waste bin.
  * The infant's legs will be kept in the flexion position and a clean diaper will be placed under them. A bottom care plan will be applied in line with the treatment plan, if necessary.
  * Tapes of the clean diaper will be fastened.
  * Hands will be washed after the procedure.
  * Data will be collected immediately before, during, immediately after and 3 minutes after the end of application.
  Arms: Experimental (Legs are flexed toward abdomen) Group

SUMMARY:
The purpose of this study is to determine the effect of diaper change position on neonatal comfort and heart rate, respiratory rate and oxygen saturation in preterm infants.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled prospective trial until reaching the entire sample group specified in the Neonatal Intensive Care Units (NICU) in a private hospital that has other branches in Istanbul.

During the data collection process, two methods will be applied to preterm infants during diaper change.

In the control group of the study, diaper change will be performed after the legs of the babies are brought to extension, and in the experimental group, the diaper change will be performed after the legs of the babies are brought closer to the abdomen by maintaining their flexion. Data on the babies' heart rate, respiratory rate, oxygen saturation and comfort level will be collected using the Premature Infant Comfort Scale before, during, immediately after and 3 minutes after the procedure.

The researchers will collect the data by using a form that questions individual characteristics and includes records of heart rate, respiratory rate and oxygen saturation and Premature Infant Comfort.

ELIGIBILITY:
Inclusion Criteria:

* The preterm infants whose
* Parents have agreed to participate in the study and have signed the informed consent form,
* Who have no congenital anomalies,
* Have no chronic illnesses,
* Have undergone Underwent no surgical procedures,
* Have no neurological symptoms,
* Have not been diagnosed with sepsis,
* Have not been sedated,
* Have not received any pharmacological analgesic method four hours before,
* Have been born between ≥28 and ≤36+6 gestational weeks or have been born earlier and are between ≥28 and ≤36+6 gestational weeks during the application, will be included.

Exclusion Criteria:

The preterm infants whose

* Parents have not agreed to participate in the study and have not signed the informed consent form,
* Who have congenital anomalies,
* Have chronic illnesses,
* Have undergone surgical procedures,
* Have neurological symptoms,
* Have been diagnosed with sepsis,
* Have been sedated,
* Have received pharmacological analgesic methods four hours before,
* Were between <28 and >36+6 gestational weeks, will be excluded.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Heart rate | Data will be collected immediately before, during, immediately after and 3 minutes after the end of application. The change in these time intervals will be assessed.
  Preterm infant will be monitored and heart rate will be monitored.
Change in Respiratory Rate | Data will be collected immediately before, during, immediately after and 3 minutes after the end of application. The change in these time intervals will be assessed.
  Preterm infant will be monitored and respiratory rate will be monitored.
Change in Oxygen Saturation | Data will be collected immediately before, during, immediately after and 3 minutes after the end of application. The change in these time intervals will be assessed.
  Preterm infant will be monitored and respiratory rate will be monitored.
Change in Comfort | Data will be collected immediately before, during, immediately after and 3 minutes after the end of application. The change in these time intervals will be assessed.
  Premature Infant Comfort Scale (PICS), which is a multidimensional scale used in evaluating comfort and pain behaviorally and psychologically. The PICS evaluates seven parameters as Alertness, Calmness/Agitation, Respiratory Status (only on mechanic ventilation support) or Crying (not evaluated because it is scored in children with spontaneous breathing), Physical Movements, Muscle Tone, Facial Gestures and Mean Heart Rate. It is a five-point likert scale in which each element is scored from one to five (from bad to good). According to the PICS, the infant's comfort is evaluated over the total score. Accordingly, 35 points signify the lowest comfort score, while seven points signify the highest comfort score. High score obtained from the scale signifies that the comfort level is low. If the total score is ≥17, this is the cut-off value of the scale. It was found that the Turkish version was a valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyngstad LT, Tandberg BS, Storm H, Ekeberg BL, Moen A. Does skin-to-skin contact reduce stress during diaper change in preterm infants? Early Hum Dev. 2014 Apr;90(4):169-72. doi: 10.1016/j.earlhumdev.2014.01.011. Epub 2014 Feb 16. PMID 24548816
- [Background] Morelius E, Hellstrom-Westas L, Carlen C, Norman E, Nelson N. Is a nappy change stressful to neonates? Early Hum Dev. 2006 Oct;82(10):669-76. doi: 10.1016/j.earlhumdev.2005.12.013. Epub 2006 Feb 28. PMID 16507341
- [Background] Kolcaba KY. Holistic comfort: operationalizing the construct as a nurse-sensitive outcome. ANS Adv Nurs Sci. 1992 Sep;15(1):1-10. doi: 10.1097/00012272-199209000-00003. PMID 1519906
- [Background] Grunau RE, Weinberg J, Whitfield MF. Neonatal procedural pain and preterm infant cortisol response to novelty at 8 months. Pediatrics. 2004 Jul;114(1):e77-84. doi: 10.1542/peds.114.1.e77. PMID 15231977
- [Background] Picheansathian W, Woragidpoonpol P, Baosoung C. Positioning of Preterm Infants for Optimal Physiological Development: a systematic review. JBI Libr Syst Rev. 2009;7(7):224-259. doi: 10.11124/01938924-200907070-00001. PMID 27820087